CLINICAL TRIAL: NCT05466695
Title: Comparing The Effect of Tadalafil 5 mg/Day to Sildenafil 25 mg/Day on Neutrophil-Lymphocyte and Platelet-Lymphocyte Ratios in Erectile Dysfunction Patients; and Comparison of Clinical Response
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed diab mohamed ramadan, Resident physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oral PDI5 and Blood components
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Erectile Dysfunction and Neutrophil Lymphocyte Ratio
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Patients will use daily tadalafil 5 mg or daily sildenafil 25 mg 4. Assessment of the grade of erectile dysfunction using international index of erectile function-5.The patients whose international Index of Erectile Function-5 (IIEF-5) scores varied between 5-7 are considered to have severe and 8-16 are considered to have moderate and 17-21 are considered to have mild erectile dysfunction.
  2. Blood sample will be obtained before and after 2 months of medical treatment to measure neutrophil-lymphocyte and platelet-lymphocyte ratios.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tadalfil group (Experimental): Patients will use daily tadalafil 5 mg for 2 months
  Interventions: Drug: Tadalafil 5mg/sildenafil 25 mg
- sildenafil group (Experimental): Patients will use daily sildenafil 25 mg for 2 months
  Interventions: Drug: Tadalafil 5mg/sildenafil 25 mg

INTERVENTIONS:
Drug: Tadalafil 5mg/sildenafil 25 mg — patients will use daily tadalafil or daily sildenafil for 2 months blood sample will be obtained before and after 2 months and also IIEF-5 score for clinical response
  Other Names: blood sample before and after 2 months of medical tratment

SUMMARY:
1- To evaluate the effect of using tadalafil 5mg/day or sildenafil 25mg/day in the treatment on these ratios and its clinical effect in erectile dysfunction patients.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is an inability to provide adequate erection to initiate or maintain any sexual activity. The ED prevalence in adult males is approximately 20%. Cardiovascular diseases, diabetes mellitus(DM), chronic systemic diseases, smoking and obesity are among the aetiology of ED .In recent years, publications indicating that active inflammatory processes cause ED are increasing. In these studies where neutrophil- lymphocyte (NLR) and platelet-lymphocyte ratios (PLR) were used as signs of inflammation, a significant relationship was found between diseases with these proportions .Neutrophil-to-lymphocyte ratio (NLR) is a simple parameter to assess easily the inflammatory status of a subject. It has proven its usefulness in the stratification of mortality in major cardiac events , as a strong prognostic factor in several types of cancers , or as a predictor and a marker of inflammatory or infectious pathologies (such is pediatric appendicitis) and postoperative complications. Through enhanced production of cytokines and expression of cellular adhesion molecules, the dysfunctional endothelium promotes inflammation within the vascular wall and sets the stage for initiation and progression of atherosclerotic lesions in both penile vasculature and in peripheral and coronary blood vessels. It has been shown that patients with vasculogenic ED have increased inflammatory activation compared to subjects without ED.There are numerous studies suggesting that phosphodiesterase-5(PDE-5) inhibitors, which are the first-line therapy of ED, might be effective in reversing generalized endothelial dysfunction. Chronic treatment restores endothelium-dependent relaxations at various sites of the vascular tree, even up to one week after cessation of the treatment . Previous studies reported a chronic effect of sildenafil and tadalafil on endothelial function and pro-inflammatory markers/mediators including intercellular and vascular cell adhesion molecules-1 (ICAM-1 and VCAM-1, respectively), high sensitivity C-reactive protein (hsCRP), and interleukin-6

ELIGIBILITY:
Inclusion Criteria:

* Male patients with mild,moderate and severe erectile dysfunction.
* Age from 25 to 60 years.

Exclusion Criteria:

* · Severe uncontrolled medical condition(DM,HTN).

  * Patients under treatment with sublingual nitrate .
  * Patients with blood diseases that affect sexual function (Leukaemia).
  * Patients using cytotoxic drugs or immunosuppressive drugs.
  * Single patient.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of tadalafil on erectile dysfunction and neutrophil-lymphocyte and platelet-lymphocyte ratios . | 2 months
  Effect of daily tadalfil 5 mg on erectile dysfunction and neutrophil-lymphocyte and platelet-lymphocyte ratios
Effect of sildenafil on erectile dysfunction and neutrophil-lymphocyte and platelet-lymphocyte ratios . | 2 months
  Effect of sildenafil 25 mg daily on erectile dysfunction and neutrophil-lymphocyte and platelet-lymphocyte ratios .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt